CLINICAL TRIAL: NCT05844826
Title: A Clinical Study To Evaluate Small Intestine Microbiome In Multiple Sclerosis (MS)
Brief Title: Evaluation of the Microbiome in Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial constraints and study recruitment phase exceeded the time allotted
Sponsor: Nimble Science Ltd. (Industry)
Collaborators: IGY Life Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REB22-1771
Record Dates: First submitted 2023-04-05; First posted 2023-05-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Participant swallows and retrieves capsule in stool. Intestinal fluid samples collected by SIMBA capsules from the MS and HC participants, along with a fecal and blood samples, will be used for gut microbiome, viral and metabolomic analysis.
  Interventions: Device: SIMBA Capsule

INTERVENTIONS:
Device: SIMBA Capsule — Participants will swallow capsule

SUMMARY:
To access the small intestinal microbiome and find abnormal microbiome/metabolome signature in luminal fluid samples from small bowel in MS compared to HC that could be used as biomarkers for MS.

DETAILED DESCRIPTION:
Participants will be swallowing the SIMBA capsule which allows for minimally-invasive sampling of the microbiome and metabolome deep in the small intestine. Researchers will use the capsule samples to access the small intestinal microbiome and find abnormal metabolomic signatures in luminal fluid samples from the small bowel in Multiple Sclerosis (MS) patients compared to healthy control.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years inclusive.
2. Have diagnosis of Multiple Sclerosis (relapsing remitting or secondary progressive for the MS cohort) or be a healthy individual living in the same household (non-MS for the healthy control cohort)
3. No antibiotics, or colon cleanses/bowel preparation in the previous 2 weeks.
4. Written informed consent

Exclusion Criteria:

1. Known to have swallowing disorders
2. Known disease which, in the investigator's opinion, would lead to intestinal stricture or obstruction with a risk of capsule non-excretion (particular diseases which would be assessed on a case-by-case basis would include, achalasia, eosinophilic esophagitis, diverticulitis, Crohn's disease, Ulcerative colitis, cancer diagnosis or treatment within the past year, or previous oesophageal, gastric, small intestinal, or colonic surgery. 3) Appendectomy or cholecystectomy more than 3 months prior to enrolment are acceptable). The main deciding factor would be history of obstructive symptoms in the previous 3 months prior to entry.
3. Use of any medications in the previous week that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics, laxatives), or acidity (PPI, H2RA); for both groups.
4. < 2 bowel movements per week (for both groups).
5. Risk or suspect of being pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
16s microbiome sequencing and LC-MS metabolomic analysis will be performed on these samples to compare gut microbiome and metabolite profiles of healthy control and diagnosed MS patients | baseline
  Comparison of luminal fluid samples from the small bowel of MS and healthy control participants will allow us to find abnormal metabolomic signatures which can be used as biomarkers for MS.
Comparison of blood samples from Multiple Sclerosis (MS) and healthy control participants for biomarkers of inflammation, as analysed using ELISA, protenomic methods, and commercially available assays. | baseline
  Comparison of blood samples from Multiple Sclerosis (MS) and healthy control participants will aid in quantification of markers of inflammation and markers of intestinal function.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camara-Lemarroy, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No